CLINICAL TRIAL: NCT05566002
Title: Artificial Intelligence-Assisted Evaluation of Pulmonary Hypertension
Acronym: AIPHY
Status: Recruiting | Type: Observational
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: AIPHY Project
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: pulmonary hypertension; pulmonary vascular disease; right heart catheterization; echocardiography; electrocardiography; chest X-ray; artificial intelligence; machine learning; deep learning; screening; diagnosis
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with pulmonary hypertension: A series of routine examinations, including chest X-ray, electrocardiography, echocardiography, etc, would be performed on consecutive patients at Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China. An RHC with an mPAP of >20 mmHg would confirm the diagnosis of PH. All these data will be collected as a source for machine learning or other artificial intelligence-assisted programs.
  Interventions: Diagnostic Test: Right heart catheterization
- Patients without pulmonary hypertension: A series of routine examinations, including chest X-ray, electrocardiography, echocardiography, etc, would be performed on consecutive patients at Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China. An RHC with an mPAP of ≤20 mmHg would confirm the absence of PH. All these data will be collected as a source for machine learning or other artificial intelligence-assisted programs.
  Interventions: Diagnostic Test: Right heart catheterization

INTERVENTIONS:
Diagnostic Test: Right heart catheterization — RHC is commonly used essential test to make gold-standard diagnosis of PH with mPAP >20 mmHg. All multimodal data from patients eligible for inclusion would be randomly assigned to development datasets (70% of the study population) to train the artificial intelligence models for the detection of PH, which would be validated and tested by other datasets (30% of the study population).

SUMMARY:
Pulmonary hypertension represents a challenging and heterogeneous condition that is associated with high mortality and morbidity if left untreated. Artificial intelligence is used to study and develop theories and methods that simulate and extend human intelligence, which is being applied in fields related to cardiovascular diseases. The study intends to combine multimodal clinical data of patients who undergo right heart catheterization at Fuwai Hospital with artificial intelligence techniques to create programs that can screen and diagnose pulmonary hypertension.

DETAILED DESCRIPTION:
Patients with pulmonary hypertension (PH) represent a challenging and heterogeneous cohort with high morbidity and mortality if left untreated. To make a definitive diagnosis of PH, one needs to conduct an invasive right heart catheterization (RHC) in order to assess the mean pulmonary artery pressure (mPAP). As PH occurs sporadically in various medical conditions, including connective tissue disease, and congenital heart disease, and presenting symptoms are non-specific, there is a need to raise the suspicion of PH early in the community. For this reason, noninvasive tools that are widely available for upfront screening would be ideal to enable timely diagnosis of PH. Transthoracic echocardiography has emerged as the mainstay for screening of PH, yet the sensitivity and specificity of this approach remain limited even in experienced hands. As high-throughput technologies advance and access to PH big data improve, it will be critical to prudently select artificial intelligence approaches for data analysis, visualization, and interpretation. By combining the multimodal clinical data (such as indicators from chest X-ray, electrocardiography, and echocardiography), this study aims to develop artificial intelligence-assisted programs to assist the screening and diagnosis of PH, and to evaluate its diagnostic accuracy for PH as compared with RHC, and to estimate whether this approach outperforms the conventional echocardiographic method.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Patients previously received chest X-ray, electrocardiography, echocardiography, other routine examinations, and RHC at the Fuwai Hospital, CAMS & PUMC, Beijing, China

Exclusion Criteria:

* Patients without RHC
* The quality of routine examinations and RHC cannot meet the requirement for further analysis
* Severe loss of results of routine examinations (chest X-ray, electrocardiography, echocardiography, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients previously received chest X-rays, electrocardiography, echocardiography, other routine examinations, and RHC at the Fuwai Hospital, CAMS & PUMC, Beijing, China.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of diagnosis by artificial intelligence-assisted algorithm | Baseline
  The investigators will calculate the area under the receiver operating characteristic curve of diagnosis by artificial intelligence-assisted algorithm and compare this index between artificial intelligence-assisted algorithm and RHC.

SECONDARY OUTCOMES:
Sensitivity of diagnosis by artificial intelligence algorithm | Baseline
  The investigators will calculate the sensitivity of diagnosis by artificial intelligence-assisted algorithm and compare this index between artificial intelligence-assisted algorithm and RHC.
Specificity of diagnosis by artificial intelligence algorithm | Baseline
  The investigators will calculate the sensitivity of diagnosis by artificial intelligence-assisted algorithm and compare this index between artificial intelligence-assisted algorithm and RHC.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD, PhD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang Z, Diao X, Huo Y, Zhao Z, Geng J, Zhao Q, Liu J, Xi Q, Xia Y, Xu O, Li X, Duan A, Zhang S, Gao L, Wang Y, Li S, Luo Q, Liu Z, Zhao W. Deep Learning-Enhanced Noninvasive Detection of Pulmonary Hypertension and Subtypes via Chest Radiographs, Validated by Catheterization. Chest. 2025 Nov;168(5):1215-1230. doi: 10.1016/j.chest.2025.06.008. Epub 2025 Jun 18. PMID 40541737
- [Derived] Zhao W, Huang Z, Diao X, Yang Z, Zhao Z, Xia Y, Zhao Q, Sun Z, Xi Q, Huo Y, Xu O, Geng J, Li X, Duan A, Zhang S, Gao L, Wang Y, Li S, Luo Q, Liu Z. Development and validation of multimodal deep learning algorithms for detecting pulmonary hypertension. NPJ Digit Med. 2025 Apr 10;8(1):198. doi: 10.1038/s41746-025-01593-3. PMID 40205021